CLINICAL TRIAL: NCT07399444
Title: A Clinical Study to Evaluate the Safety, Tolerability, and Efficacy of the LVIVO-TaVec400 Product in the Treatment of Relapsed/Refractory Multiple Myeloma
Brief Title: A Clinical Study to Evaluate LVIVO-TaVec400 for the Treatment of Relapsed/Refractory Multiple Myeloma（LB2505-0001）
Acronym: LB2505-0001
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Nanjing Legend Biotech Co. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025143
Record Dates: First submitted 2026-01-25; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Multiple Myeloma (MM)
Keywords: Relapsed/Refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LVIVO-TaVec400 product (Experimental): Each subject will be given a single-dose LVIVO-TaVec400 product infusion at each dose level
  Interventions: Biological: LVIVO-TaVec400 product

INTERVENTIONS:
Biological: LVIVO-TaVec400 product — Prior to infusion of the LVIVO-TaVec400 product, subjects will receive bridging therapy if needed.

SUMMARY:
This is a prospective, single-arm, open-label dose-escalation clinical study to evaluate LVIVO-TaVec400 in the treatment of relapsed/refractory multiple myeloma.

DETAILED DESCRIPTION:
This is a prospective, single-arm, open-label dose-escalation and dose-expansion study, designed to evaluate the safety, tolerability, anti-tumor efficacy profile, and pharmacokinetic characteristics of the LVIVO-TaVec400 in subjects with relapsed/refractory multiple myeloma who have failed at least 3 lines of prior standard therapies. The subject who meet the defined eligibility criteria will be enrolled with a core study period of approximately 2 years, including the screening, bridging therapy(if needed), treatment, and follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily participate in clinical studies; Fully informed of this study and signed informed consent; Informed consent form must be obtained prior to initiation of any study-related tests or procedures that are not part of the standard treatment for the subject's disease; Good compliance and cooperation with follow-up.
2. Age ≥ 18 years.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Has measurable lesions
5. Relapsed and/or refractory multiple myeloma
6. Life expectancy≥ 3 months
7. Clinical laboratory values meet screening visit criteria
8. Adequate organ function.

Exclusion Criteria:

1. Prior antitumor therapy with insufficient washout period ;
2. Patients who are positive for hepatitis B surface antigen (HBsAg), hepatitis B virus deoxyribonucleic acid (HBV DNA), hepatitis C antibody (HCV-Ab), hepatitis C virus ribonucleic acid (HCV RNA), and human immunodeficiency virus antibody (HIV-Ab).
3. Those who have experienced life-threatening allergic reactions, hypersensitivity reactions or intolerances to the excipients and related additives of the investigational drug; or those with a previous history of severe allergic reactions (such as hypersensitivity reactions, or those for whom the investigator assesses the need to use glucocorticoids to prevent severe immune-related reactions such as allergic reactions).
4. Any condition deemed by the investigator as rendering the subject unsuitable for participation in this study.
5. Also enrolled in other clinical studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2028-07-10 (Estimated); Study Completion 2030-05-10 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) incidence rate and the incidence, severity and type of adverse events (TEAEs) during treatment. | Through study completion, an average of 2 years after LVIVO-TaVec400 infusion (Day 1)
Determine the recommended dose (RP2D) for the treatment of this research formulation in the Phase II clinical trial. | Through study completion, an average of 2 years after LVIVO-TaVec400 infusion (Day 1)
Pharmacokinetics in peripheral blood | Through study completion, an average of 2 years after LVIVO-TaVec400 infusion (Day 1)
  CAR positive T cells and CAR transgene percentage of in peripheral blood after LVIVO-TaVec400 infusion
Pharmacokinetics in bone marrow | Through study completion, an average of 2 years after LVIVO-TaVec400 infusion (Day 1)
  CAR positive T cells and CAR transgene percentage of in bone marrow after LVIVO-TaVec400 infusion

CONTACTS AND LOCATIONS:
Overall Officials: Lugui Qiu, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (6):
- China (6):
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Beijing GoBroad Boren Hospital, Beijing
  - Institute of Hematology & Blood Diseases Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: No